CLINICAL TRIAL: NCT01153490
Title: Improving Substance Use and Clinical Outcomes in Heavy Cannabis Users With Quetiapine
Acronym: CD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Raphael Braga, Perioperative Assistant, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-159B
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Cannabis Dependence
Keywords: Quetiapine; Psychotic experiences; Cannabis dependence; Craving; Mood; Substance use
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Behavioral Intervention
- Quetiapine ER (Active Comparator)
  Interventions: Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Substance-related

SUMMARY:
Cannabis is the most used illicit substance in the United States. Previous studies suggest that atypical antipsychotics decrease the frequency and the amount of substance use in subjects with and without psychotic illness. So far, there are no controlled studies assessing the effectiveness of atypical antipsychotics for decreasing cannabis and other substance use in individuals with cannabis use disorders. The investigators postulate that the atypical antipsychotic quetiapine ER is an effective agent for improving substance use outcomes in subjects with cannabis use disorders. In this pilot study, the investigators will test this hypothesis in heavy cannabis users (i.e., individuals who are cannabis dependent and smoke three times or more per week). Because 50% of these heavy cannabis users report histories of psychotic experiences (i.e., attenuated positive symptoms) while smoking and are at risk for recurring psychotic symptoms, the investigators will focus this pilot clinical trial on this subgroup of cannabis users in order to increase the risk/benefit ratio of this study and target a population that may also benefit from the antipsychotic effect of quetiapine ER. Considering the lack of controlled studies assessing the efficacy of atypical antipsychotics in heavy cannabis users, assessing the effectiveness of an atypical antipsychotic medication on substance use and clinical outcomes in this population is critical for improving the prognosis of these individuals.

Thus, the aims of this randomized, double-blind, placebo-controlled study are to assess the efficacy of an atypical antipsychotic (quetiapine ER) in 120 subjects with cannabis dependence, a recent history (within a year) of attenuated psychotic symptoms, and using cannabis 3 times or more per week for: (1) decreasing the use of cannabis and other substances; and (2) preventing the recurrence of psychotic experiences. The investigators will also assess the effects of quetiapine ER on craving and mood, and its tolerability. This project will be a 12-week, randomized, double-blind, placebo-controlled study with quetiapine ER and it will include a comprehensive assessment of symptoms, substance use, and side effects.

This study will benefit the field by providing unique data on the relative efficacy and tolerability of treatment with atypical antipsychotics in heavy cannabis users with a vulnerability to psychosis. This study will be the basis for future studies assessing the long-term efficacy and tolerability of atypical antipsychotics in individuals with cannabis use disorders.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-defined diagnosis of cannabis dependence (304.30) assessed with the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I/P) (First 1998))
* one or more attenuated positive symptoms with a score 3 ('moderate'), 4 ('moderate severe'), or 5 ('severe but not psychotic') during the past year assessed with the Structured Interview for Prodromal Syndromes (SIPS) and the Scale of Prodromal Symptoms (SOPS) (McGlashan et al, 2001)
* lifetime treatment with antipsychotic medication less than 2 weeks
* cannabis use for more than one year
* cannabis use three or more days per week on average for the past 3 months
* aged 18 to 65
* competent and willing to sign informed consent
* for women, a negative urine pregnancy test and agreement to use a medically accepted method of birth control during the study.

Exclusion Criteria:

* DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, a psychotic disorder due to a general medical condition, psychosis NOS, delusional disorder, brief psychotic disorder, shared psychotic disorder, or a mood disorder (major depression or bipolar) with psychotic features assessed with the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I/P) (First 1998)
* DSM-IV diagnosis of any psychoactive substance dependence other than cannabis or nicotine
* being in an environment with no access to cannabis (e.g., hospitalization, residential treatment, jail, ..) for more than one week during the past three months preceding study entry
* serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain
* use of medications that have an effect on monoamines (e.g., antidepressants
* severe medical or physical illnesses
* criteria of the National Cholesterol Education Program (NCEP) for a metabolic syndrome (Expert panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults, 2001)
* medical condition that requires treatment with a medication that has psychotropic effects
* significant risk of suicidal or homicidal behavior
* cognitive or language limitations, or any other factor that would preclude subjects providing informed consent or participating in study procedures
* treatment with medications for addiction
* treatment with medication having a risk of addiction (e.g., benzodiazepines, barbiturates)
* history of treatment resistance to quetiapine ER
* medical contraindications to quetiapine ER
* hypersensitivity to quetiapine ER or any of its component
* for women, pregnant, breastfeeding, or intention to become pregnant during the study timeframe

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-10-22 (Actual); Primary Completion 2012-08-06 (Actual); Study Completion 2012-08-06 (Actual)

PRIMARY OUTCOMES:
Frequency/amount of substance use | 12 weeks
  frequency and amount of cannabis and other substance use will be recorded with the Timeline Follow-Back Method.
Psychotic symptoms | 12 weeks
  Psychotic symptoms wil be assessed with the Structured Interview for Prodromal Symptoms and the Brief Psychiatric Rating Scale.

SECONDARY OUTCOMES:
Craving | 12 weeks
  Craving will be assessed with the Marijuana Craving Questionnaire and a Visual Analog Craving Scale
Mood symptoms | 12 weeks
  Mood symptoms will be assessed with the Hamilton Depression Rating Scale
Adverse events | 12 weeks
  Adverse events will be assessed with the Systematic Assessment for Treatment Emergent Events interview, Simpson-Angus Scale for Extrapyramidal Symptoms, the Abnormal Involuntary Movement Scale, the Barnes Akathisia Scale, and blood tests (fasting glucose, insulin and lipid profile tests)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Sevy, M.D., MBA, Principal Investigator — Feinstein Institute for Medical Research
Locations (2):
- United States (2):
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - General Clinical Research Center, Manhasset, New York